CLINICAL TRIAL: NCT06365255
Title: National Epidemiological Study of the Possible Impact of Stress on Glycaemic Control in Patients With Type 1 Diabetes
Acronym: EPISTRESS2
Status: Completed | Type: Observational
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01453-40
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Type 1
Keywords: Stress; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires — filling in questionnaires

SUMMARY:
The EPISTRESS2 study is a one-off cross-sectional epidemiological survey, carried out via an online form in patients with type 1 diabetes followed up by participating investigating centres.

In type 1 diabetes (T1DM), studies on stress and its impact on glycaemia have led to ambiguous results, mainly because there are no solid epidemiological or experimental data in the literature. The aim of this study was to assess the impact of perceived stress on blood glucose levels in a population of subjects with T1DM at 10 national centres.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes;
* Do not have a psychiatric pathology;
* At least 18 years old;
* Affiliated to the Social Security;
* Having read the non-opposition form and not objecting to it.

Exclusion Criteria:

* Patient who has declared his opposition using the electronic non-opposition form
* Patient with type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To study the impact of stress on glycaemia, we chose to conduct an epidemiological study in France on a population of type 1 diabetic patients (T1DM).
  Many patients frequently and systematically cite stress as a frequent cause, or even the main cause, of the deterioration in their glycaemic control.
Sampling Method: Non-Probability Sample
Enrollment: 1344 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the characterisation of 4 profiles of patients with type 1 diabetes on insulin pumps. | 30 minutes
  Questionnaire for Assessing the Impact of Stress on Blood Sugar Levels. This questionnaire was designed and developed by CERITD to assess the impact of perceived stress on blood glucose levels in T1DM patients.

SECONDARY OUTCOMES:
Identify sub-populations of patients who feel stressed | 30 minutes
  * Identify and profile a sub-population of patients whose blood glucose levels rise in response to stress
  * Identify and profile a sub-population of patients whose blood glucose levels decrease in response to stress
  Questionnaire for Assessing the Impact of Stress on Blood Sugar Levels
Establish and categorise the different stress factors | 30 minutes
  Cungi brief stress evaluation scales The Cungi 1 scale is composed of 8 items. This questionnaire assesses patient stressors.
  The maximum score is 48, the minimum score is 8. A high score reflects a large number of stressors
  The Cungi 2 scale is composed of 11 items. This questionnaire assesses the patient's sensitivity to stress.
  The maximum score is 66, the minimum score is 11. A high score reflects a high senstivity of stress.
Establishing a relationship between personality type and the impact of stress | 30 minutes
  State-Trait Anxiety Inventory (STAI) questionnaire. The STAI-Y1 is composed of 20 items. This questionnaire assesses how the patient feels at the present moment. Patients are asked to score each question on a four-point scale (from 1 - corresponding to "not at all" to 4 - "much")
  The STAI-Y2 is composed of 20 items. This questionnaire assesses how the patient feels in general.
  Patients are asked to answer each question on a four-point scale (from 1 - corresponding to "almost never" to 4 - "almost always").
Evaluation of the quality of life score obtained according to the 4 profiles and/or personalities | 30 minutes
  EQ-5D-5L (European Quality of Life 5 Dimensions) questionnaire The EQ-5D-5L assesses five health dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is rated on five levels of severity. The levels of severity for each dimension ranges from no problems (1) to extreme problems/unable to perform (5)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Franc, MD, Principal Investigator — Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète
Locations (11):
- France (11):
  - Angers University Hospital, Angers
  - Avignon Hospital, Avignon
  - St André Hospital, Bordeaux
  - Brest University Hospital, Brest
  - Dijon University Hospital, Dijon
  - CERITD, Évry
  - Grenoble University Hospital, Grenoble
  - Lille University Hospital, Lille
  - APHM- La Conception Hospital, Marseille
  - Private practice in endocrinology and metabolic diseases, Mérignac
  - Srasbourg University Hospital, Strasbourg